CLINICAL TRIAL: NCT03627767
Title: A PHASE 3 RANDOMIZED WITHDRAWAL, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTI-CENTER STUDY INVESTIGATING THE EFFICACY AND SAFETY OF PF-04965842 IN SUBJECTS AGED 12 YEARS AND OVER, WITH MODERATE TO SEVERE ATOPIC DERMATITIS WITH THE OPTION OF RESCUE TREATMENT IN FLARING SUBJECTS
Brief Title: Study to Investigate Efficacy and Safety of PF-04965842 in Subjects Aged 12 Years and Over With Moderate to Severe Atopic Dermatitis With the Option of Rescue Treatment in Flaring Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7451014; JADE REGIMEN (Other: Alias Study Number); 2018-000501-23 (EudraCT Number); REGIMEN (Other: Alias Study Number)
Record Dates: First submitted 2018-05-29; First posted 2018-08-13 (Actual); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Dermatitis; Dermatitis, Atopic; Eczema; Skin Diseases; Skin Diseases, Genetic; Genetic Diseases, Inborn; Skin Diseases, Eczematous; Hypersensitivity; Hypersensitivity, Immediate; Immune System Diseases
Keywords: atopic dermatitis; atopic eczema; eczema; JAK; janus kinase
MeSH Terms: conditions — Dermatitis; Dermatitis, Atopic; Eczema; Skin Diseases; Skin Diseases, Genetic; Genetic Diseases, Inborn; Skin Diseases, Eczematous; Hypersensitivity; Hypersensitivity, Immediate; Immune System Diseases | interventions — abrocitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PF-04965842 100 mg QD (Experimental): Double-blind randomized treatment following open label run-in period.
  Interventions: Drug: PF-04965842 100 mg
- PF-04965842 200 mg QD (Experimental): Double-blind randomized treatment following open label run-in period.
  Interventions: Drug: PF-04965842 200 mg
- Placebo QD (Placebo Comparator): Double-blind randomized treatment following open label run-in period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04965842 100 mg — PF-04965842 100 mg, administered as two tablets to be taken orally once daily for 40 weeks
  Other Names: Abrocitinib
  Arms: PF-04965842 100 mg QD
Drug: PF-04965842 200 mg — PF-04965842 200 mg, administered as two tablets to be taken orally once daily for 40 weeks
  Other Names: Abrocitinib
  Arms: PF-04965842 200 mg QD
Drug: Placebo — Placebo, administered as two tablets to be taken orally once daily for 40 weeks
  Arms: Placebo QD

SUMMARY:
B7451014 is a Phase 3 study to investigate PF-04965842 in patients aged 12 years and over with a minimum body weight of 40 kg who have moderate to severe atopic dermatitis. Subjects responding well to an initial open-label 12 week treatment of PF-04965842 (200 mg) taken orally once daily (QD) will be identified and randomized in a double-blind manner to receive 200 mg QD PF-04965842, 100 mg QD PF-04965842, or QD placebo. Efficacy and safety of 2 doses of PF-04965842 will be evaluated relative to placebo over 40 weeks. Subjects experiencing significant worsening of their symptoms, i.e., protocol-defined flare, enter 12 weeks rescue treatment and receive 200 mg PF-04965842 together with a marketed topical medicine. Eligible patients will have the option to enter a long-term extension study after completing the initial 12 week treatment, the 12 week rescue treatment, and the 40 week blinded treatment.

DETAILED DESCRIPTION:
Responder criteria for randomization at week 12 are defined as a) achieving an IGA of clear (0) or almost clear (1) (on a 5 point scale), b) a reduction from IGA baseline of 2 or more points, and c) reaching an EASI-75 response compared to baseline. Flare requiring rescue treatment is defined as a loss of at least 50% of the EASI response at Week 12 and an IGA score of 2 or higher.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older with a minimum body weight of 40 kg
* Diagnosis of atopic dermatitis (AD) for at least 1 year and current status of moderate to severe disease (>= the following scores: BSA10%, IGA 3, EASI 16, Pruritus NRS 4)
* Recent history of inadequate response or inability to tolerate topical AD treatments or require systemic treatments for AD control

Exclusion Criteria:

* Unwilling to discontinue current AD medications prior to the study or require treatment with prohibited medications during the study
* Prior treatment with JAK inhibitors
* Other active nonAD inflammatory skin diseases or conditions affecting skin
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, Q wave interval abnormalities, current or history of certain infections, cancer, lymphoproliferative disorders and other medical conditions at the discretion of the investigator
* Pregnant or breastfeeding women, or women of childbearing potential who are unwilling to use contraception

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1235 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (235):
- United States (52):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - University of Alabama at Birmingham, Dermatology at the Whitaker Clinic, Birmingham, Alabama
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - Tien Q Nguyen MD Inc dba First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Beach Allergy and Asthma Specialty Group, A Medical Corporation, Long Beach, California
  - Dermatology Specialists, Inc., Oceanside, California
  - University of California San Diego, San Diego, California
  - San Luis Dermatology and Laser Clinic, San Luis Obispo, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - Mosaic Dermatology, Santa Monica, California
  - Bay Pines VAHCS, Bay Pines, Florida
  - Skin Care Research, LLC, Boca Raton, Florida
  - Skin Research Institute, Coral Gables, Florida
  - Baumann Cosmetic and Research Institute, Miami, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - USF Asthma, Allergy & Immunology Clinical Research Unit, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Dermatologic Surgery Specialists, PC, Macon, Georgia
  - Midwest Allergy Sinus Asthma, SC, Normal, Illinois
  - NorthShore University HealthSystem Dermatology Clinical Trials Unit, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Ds Research, New Albany, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Kansas City Dermatology, P.A., Overland Park, Kansas
  - DXP Imaging, Louisville, Kentucky
  - Skin Sciences PLLC, Louisville, Kentucky
  - Qualmedica Research, LLC, Owensboro, Kentucky
  - Owensboro Dermatology Associates, Owensboro, Kentucky
  - Meridian Clinical Research, LLC, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Saint Louis University Dermatology, St Louis, Missouri
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Juva Skin and Laser Center, New York, New York
  - UR Dermatology at College Town, Rochester, New York
  - M3 - Wake Research, Inc., Raleigh, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Newton Clinical Research, Oklahoma City, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - Paddington Testing Co, Inc., Philadelphia, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Dermatology Treatment & Research Center, PA, Dallas, Texas
  - Innovate Research, LLC, Fort Worth, Texas
  - The University of Texas Health Science Center Houston, Houston, Texas
  - Ventavia Research Group Hurst, Hurst, Texas
  - Virginia Clinical Research, Inc, Norfolk, Virginia
  - Dermatology Associates of Seattle, Seattle, Washington
  - Dermatology Specialists of Spokane, Spokane, Washington
- Argentina (6):
  - Framingham Centro Medico, La Plata, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Servicio de Investigacion de Patolog-ias Alergicas del Instituto ABC, Rosario, Santa Fe Province
  - CINME Centro de Investigaciones Metabolicas, C.a.b.a.
  - Buenos Aires Skin, C.a.b.a.
  - Psoriahue Medicina Interdisciplinaria, C.a.b.a
- Belgium (3):
  - University Hospital Brussels, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital Antwerp, Edegem
- Brazil (7):
  - CETI - Centro de Estudos em Terapias Inovadoras LTDA., Curitiba, Paraná
  - Instituto de Dermatologia e Estética do Brasil LTDA, Rio de Janeiro, Rio de Janeiro
  - Hospital De Clinicas De Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Associacao dos Funcionarios Públicos do Estado do Rio Grande do Sul - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Pesquisare Saude S/S Ltda, Santo André, São Paulo
  - Fundacao do ABC - Faculdade de Medicina do ABC, Santo André, São Paulo
  - IBPClin Pesquisa Clinica, Rio de Janeiro
- Bulgaria (7):
  - MC Asklepii" OOD, Dupnitsa
  - MHAT "Dr. Tota Venkova" AD, Gabrovo
  - "Center of skin-venereal diseases" EOOD, Sofia, Sofia
  - "DCC Fokus-5-Medical Establishment for OutpatientCare"EOOD, Sofia
  - "Mc Sinexus Sofia" Eood, Sofia
  - ACIBADEM City Clinic Diagnostic-Consultative Center EOOD, Sofia
  - "ACIBADEM City Clinic Medical Center Varna" EOOD, Varna
- Canada (16):
  - Dermatology Research Institute, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - Alberta Dermasurgery Center, Edmonton, Alberta
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Karma Clinical Trials, Inc., St. John's, Newfoundland and Labrador
  - CCA Medical Research, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - Dermatology Ottawa Research Centre, Ottawa, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - Office of Dr. Paul Adam, Scarborough Village, Ontario
  - AvantDerm, Toronto, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - XLR8 Medical Research Inc., Windsor, Ontario
  - Centre de Recherche Dermatologique du Quebec Metropolitain (CRDQ), Québec, Quebec
- Chile (4):
  - Centro Medico SkinMed Limitada, Santiago, Santiago Metropolitan
  - Clinica Dermacross S.A., Santiago, Santiago Metropolitan
  - Hospital Clinico Universidad de Chile, Santiago, Santiago Metropolitan
  - Centro Internacional de Estudios Clinicos - CIEC, Santiago, Santiago Metropolitan
- China (20):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Army Medical University, PLA, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - Tongji Hospital, Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital With Nanjing University, Nanjing, Jiangsu
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - Jinan Central Hospital, Jinan, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Dermatological Department, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine/Dermatology and STD Dept, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine/Dermatology Dept, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital/Dermatology Department, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Peking University First Hospital, Beijing
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai Dermatology Hospital, Shanghai
- Germany (18):
  - Charite - Universitaetsmedizin Berlin, Klinik fuer Dermatologie, Venerologie und Allergologie, Berlin
  - Hautzentrum Friedrichshain Studien, Berlin
  - Rothhaar Studien GmbH, Berlin
  - Klinikum Bielefeld Rosenhoehe, Bielefeld
  - Universitaetsklinikum Bonn, Bonn
  - Universitaetsklinikum Carl Gustav Carus der Technischen Universitaet Dresden, Dresden
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Essen, Essen
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Universitätsklinikum und Poliklinik für Dermatologie und Venerologie, Halle
  - Klinische Forschung Hamburg GmbH, Hamburg
  - TFS Trial Form Support GmbH, Hamburg
  - Katholisches Kinderkrankenhaus Wilhemstift, Hamburg
  - MENSINGDERMA research GmbH, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Praxis Dr. med. Beate Schwarz, Langenau
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
  - Hautaerztliche Gemeinschaftspraxis Dres. Leitz und Kollegen, Stuttgart
- Israel (5):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - AOU Policlinico Sant'Orsola Malpighi, Bologna, BO
  - Universita' degli Studi G. D'Annunzio -CeSi-MeT, Chieti, CH
  - IFO Istituto Dermatologico San Gallicano IRCCS,, Roma, RM
  - Ospedale Cristo Re, Roma, ROME
  - Azienda Ospedaliero Universitaria San Martino di Genova, Genova
  - Ospedale Luigi Sacco, Milan
  - Prof. Giovanni Pellacani AOU Policlinico di Modena Struttura Complessa di Dermatologia, Modena
  - Universita del Sacro Cuore, Policlinico Agostino Gemelli, Istituto Di Dermatologia, Rome
- Latvia (4):
  - Riga 1st Hospital, Clinic of Dermatology and STD, Riga
  - Health and Aesthetics Ltd, Riga
  - Health Centre 4 Ltd, Dermatology Clinics, Riga
  - Outpatient Clinic Of Ventspils, Ventspils
- Mexico (6):
  - Arke Estudios Clinicos S.A. de C.V., Cuauhtémoc, Mexico City
  - JM Research SC, Cuernavaca, Morelos
  - Centro de Dermatologia de Monterrey, Monterrey, Nuevo León
  - Phylasis Clinicas Research S. de R.L. de C.V., Cuautitlán Izcalli, State of Mexico
  - Derma Norte del Bajio S.C, Aguascalientes
  - Centro de Investigacion Integral Medivest S.C., Chihuahua City
- Universitair Medisch Centrum (UMC) Utrecht, Utrecht, Netherlands
- Poland (28):
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz
  - Centrum Medyczne SENSEMED, Chorzów
  - Copernicus Podmiot Leczniczy Sp. z.o.o., Oddzial Dermatologii, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Klinika Dermatologii, Wenerologii i Alergologii, Gdansk
  - Silmedic Sp. z o.o., Oddzial w Katowicach, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Pro Familia Altera Sp. z o.o., Katowice
  - Malopolskie Centrum Kliniczne, Krakow
  - Centrum Badan Klinicznych JCI, Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - NZOZ "DERMED" Centrum Medyczne Sp. z o.o. - Oddzial w Lodzi, Lodz
  - O?rodek Bada? Klinicznych Appletreeclinics, Lodz
  - Dermoklinika-Centrum Medyczne s.c., Lodz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Laser Clinic S.C. dr Tomasz Kochanowski dr Andrzej Krolicki, Szczecin
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp. z o.o., Tarnów
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administracji w Warszawie, Warsaw
  - RCMed Oddzial Warszawa, Warsaw
  - Klinika Ambroziak Sp. z o.o., Warsaw
  - ETG Warszawa, Warsaw
  - Wojskowy Instytut Medyczny, Klinika Dermatologiczna, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
  - Lukasz Matusiak "4Health', Wroclaw
  - Kliniczny Oddzial Chorob Wewnetrznych, Dermatologii i Alergologii, Zabrze
- Romania (3):
  - SC Centrul Medical de Diagnostic si Tratament Ambulator Neomed SRL, Brasov, JUD. Brasov
  - Cabinet Medical de Dermatovenerologie Prof. Dr. Orasan Remus Ioan, Cluj-Napoca, JUD. CLUJ
  - SC Delta Health Care SRL, Bucharest
- Russia (15):
  - SBIH "Chelyabinsk Regional Clinical Dermatovenerology dispensary", Chelyabinsk
  - Limited Liability Company "Medical Center "Rheuma-Med", Kemerovo
  - Clinic of FSBEI HE Kirov SMU MOH Russia, Kirov
  - FSBI "State Research Centre of Dermatovenereology and Cosmetology" MoH RF, Moscow
  - NRC Institute of Immunology FMBA of Russia, Moscow
  - SBI RR "Skin and Venereal Dispensary", Rostov-on-Don
  - SBI RR "Regional Clinical Skin and Veneral Dispensary", Ryazan
  - LLC "Pierre Wolkenstein Clinic of Skin Diseases", Saint Petersburg
  - Vitiligo center, Saint Petersburg
  - SPb SBIH "Dermatovenerologic Dispensary #10 - Clinic of dermatology and venerology", Saint Petersburg
  - FSBEI HE "St. Petersburg State Pediatric Medical University" MoH RF, Saint Petersburg
  - Limited Liability Company "Sanavita", Saint Petersburg
  - Medical Research Institute, LLC, Saint Petersburg
  - FSBEI HE I.P.Pavlov SPbSMU MOH Russia, Saint Petersburg
  - RSBIH "Smolensk Regional Clinical Hospital", Smolensk
- Serbia (3):
  - Military Medical Academy, Belgrade
  - Clinical Centre Nis, Niš
  - General Hospital Pancevo, Pančevo
- Slovakia (8):
  - Fakultna Nemocnica s Poliklinikou F. D. Roosevelta Banska Bystrica, Banská Bystrica
  - Narodny ustav detskych chorob, Detska dermatovenerologicka klinika LF UK a NUDCH, Bratislava
  - BeneDerma s.r.o., Bratislava
  - Derma therapy spol. s.r.o, Dermatovenerologicka ambulancia, Bratislava
  - Nemocnica Kosice-Saca, a.s., 1. sukromna nemocnica, Kozna ambulancia, Kosice-Saca
  - Pedi-Derma s.r.o., Dermatovenerologicka ambulancia, Košice
  - Derma-beauty, s.r.o., Dermatovenerologicka ambulancia, Nitra
  - SANARE spol. s.r.o., Dermatovenerologicka ambulancia, Svidník
- Spain (15):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital del Nino Jesus, Madrid
  - Hospital Universitario Virgen de la Macarena, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario y Politecnico La Fe, Valencia
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Paller AS, Eichenfield LF, Irvine AD, Flohr C, Wollenberg A, Barbarot S, Bangert C, Spergel JM, Selfridge A, Biswas P, Fan H, Alderfer J, Watkins M, Koppensteiner H. Integrated Efficacy and Safety Analysis of Abrocitinib in Adolescents With Moderate-to-Severe Atopic Dermatitis. Allergy. 2025 Aug;80(8):2213-2224. doi: 10.1111/all.16512. Epub 2025 Mar 3. PMID 40028832
- [Derived] Armstrong AW, Alexis AF, Blauvelt A, Silverberg JI, Feeney C, Levenberg M, Chan G, Zhang F, Fostvedt L. Predicting Abrocitinib Efficacy at Week 12 Based on Clinical Response at Week 4: A Post Hoc Analysis of Four Randomized Studies in Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Jul;14(7):1849-1861. doi: 10.1007/s13555-024-01183-3. Epub 2024 Jun 19. PMID 38896380
- [Derived] Flohr C, Cork MJ, Ardern-Jones MR, Eichenfield LF, Barbarot S, Feeney C, Rojo R, Lazariciu I, Nesnas J. Efficacy and safety of abrocitinib monotherapy in adolescents and adults: a post hoc analysis of the phase 3 JAK1 atopic dermatitis efficacy and safety (JADE) REGIMEN clinical trial. J Dermatolog Treat. 2023 Dec;34(1):2200866. doi: 10.1080/09546634.2023.2200866. PMID 37036183
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population pharmacokinetic-pharmacodynamic modelling of platelet time-courses following administration of abrocitinib. Br J Clin Pharmacol. 2022 Aug;88(8):3856-3871. doi: 10.1111/bcp.15334. Epub 2022 Apr 11. PMID 35342978
- [Derived] Simpson EL, Silverberg JI, Nosbaum A, Winthrop KL, Guttman-Yassky E, Hoffmeister KM, Egeberg A, Valdez H, Zhang M, Farooqui SA, Romero W, Thorpe AJ, Rojo R, Johnson S. Integrated Safety Analysis of Abrocitinib for the Treatment of Moderate-to-Severe Atopic Dermatitis From the Phase II and Phase III Clinical Trial Program. Am J Clin Dermatol. 2021 Sep;22(5):693-707. doi: 10.1007/s40257-021-00618-3. Epub 2021 Aug 18. PMID 34406619
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 1235 participants were enrolled in 236 sites in 21 countries. Study started from 11 June 2018 and completed on 07 October 2020.
Pre-assignment Details: Study Baseline: was defined as the last observation collected on or prior to Day 1 (first dose day) of study treatment. Randomization Baseline: was defined as the last observation collected between last dose of run-in treatment and Day 1 (first dose day) of randomized treatment. Rescue Baseline: was defined as the last observation collected between last dose of blinded treatment and Day 1 (first dose day) of rescue treatment.
Groups:
- PF-04965842 200 mg OL: Participants received 12 weeks induction treatment of 200 milligram (mg) oral tablets (each tablet of 100 mg) PF-04965842 once daily (QD) during an OL run-in period. Responders at the end of the 12-week OL run-in period entered the 40 week, double-blind (DB), maintenance treatment period. Responder criteria was defined as a) achieving an Investigator's Global Assessment (IGA) of clear (0) or almost clear (1) (on a 5-point scale), b) a reduction from IGA baseline of greater than or equal to (>= 2) points, and c) reaching an Eczema Area and Severity Index (EASI)-75 response compared to baseline score. Baseline score was the IGA score and EASI score obtained prior to dosing on Day 1. Non-responders had a choice to enroll into the PF-04965842 Long Term Extension (LTE) study B7451015 (NCT03422822) otherwise, they were permanently discontinued from treatment and were followed-up for 4-week in this study.
- PF-04965842 200 mg OL to Placebo DB: Responders from OL run-in period received two placebo tablets matched to PF-04965842 orally QD during DB period for up to 40 weeks. Participants who met the protocol defined flare criteria entered in open-label rescue period (RP). Flare was define as a loss of at least 50 percent (%) of the EASI response at Week 12 and had an IGA score of 2 or higher. Participants who did not met the flare criteria had a choice to enroll into the LTE study, otherwise they were permanently discontinued from treatment and were followed-up for 4-week in this study.
- PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB: Responders from open-label run-in period received a tablet of 100 mg PF-04965842 and a tablet of matching placebo orally QD during DB period for up to 40 weeks. Participants who met the protocol defined flare criteria entered in open-label rescue period. Flare was define as a loss of at least 50% of the EASI response at Week 12 and had an IGA score of 2 or higher. Participants who did not met the flare criteria had a choice to enroll into the LTE study, otherwise they were permanently discontinued from treatment and were followed-up for 4-week in this study.
- PF-04965842 200 mg OL to PF-04965842 200 mg DB: Responders from open-label run-in period received 200 mg PF-04965842 (2 tablets of 100 mg each) orally QD during DB period for up to 40 weeks. Participants who met the protocol defined flare criteria entered in open-label rescue period. Flare was define as a loss of at least 50% of the EASI response at Week 12 and had an IGA score of 2 or higher. Participants who did not met the flare criteria had a choice to enroll into the LTE study, otherwise they were permanently discontinued from treatment and were followed-up for 4-week in this study.
- PF-04965842 200 mg Rescue Period: Participants who met the protocol defined flare criteria in DB period received 200 mg PF-04965842 (2 tablets of 100 mg each) orally QD during open-label Rescue Period for up to 12 weeks. After completing the 12-week rescue period, participants had the choice to enter the LTE study B7451015 (NCT03422822), if eligible. Participants who discontinued early from treatment, or who were otherwise ineligible for the LTE study, were followed-up for 4 week in this study.
Period: Open-label (OL) Run-in Period (12 Weeks)
Arm/Group | PF-04965842 200 mg OL | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB | PF-04965842 200 mg Rescue Period
Started | 1235 | 0 | 0 | 0 | 0
Treated | 1233 | 0 | 0 | 0 | 0
Completed | 798 | 0 | 0 | 0 | 0
Not Completed | 437 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 48 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 315 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 13 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 11 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 40 | 0 | 0 | 0 | 0
Not completed — Medication Error Without Associated Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal By Parent/Guardian | 2 | 0 | 0 | 0 | 0
Not completed — Other | 4 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 2 | 0 | 0 | 0 | 0
Period: Double-blind Treatment Period (40 Weeks)
Arm/Group | PF-04965842 200 mg OL | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB | PF-04965842 200 mg Rescue Period
Started | 0 (Participants did not enter into the DB period.) | 267 (Participants who met the pre-defined criteria for DB.) | 265 (Participants who met the pre-defined criteria for DB.) | 266 (Participants who met the pre-defined criteria for DB.) | 0
Participants Entered Rescue Period | 0 | 208 | 109 | 44 | 0
Completed After Entering Rescue Period | 0 | 201 | 99 | 41 | 0
Completed Without Entering Rescue Period | 0 | 43 | 134 | 187 | 0
Completed | 0 | 251 (208 entered RP+43 completed study in DB period) | 243 (109 entered RP+134 completed study in DB period) | 231 (44 entered RP+187 completed study in DB period) | 0
Not Completed | 0 | 16 | 22 | 35 | 0
Not completed — Adverse Event | 0 | 6 | 7 | 19 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 3 | 0
Not completed — Protocol Violation | 0 | 1 | 5 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 9 | 6 | 10 | 0
Not completed — Withdrawal By Parent/Guardian | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 1 | 0
Period: Open-label Rescue Period (12 Weeks)
Arm/Group | PF-04965842 200 mg OL | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB | PF-04965842 200 mg Rescue Period
Started | 0 | 0 (Participants did not enter into the OL- Rescue Period.) | 0 (Participants did not enter into the OL- Rescue Period.) | 0 (Participants did not enter into the OL- Rescue Period.) | 361 (Participants who met the pre-defined criteria for OL- Rescue Period.)
Met Protocol-defined Flare Criteria | 0 | 0 | 0 | 0 | 351
Completed | 0 | 0 | 0 | 0 | 341
Not Completed | 0 | 0 | 0 | 0 | 20
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 9
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 9
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set-randomized (FAS-RA) included as all participants who were randomized at Week 12 and received at least 1 dose of study medication within Double-blind (DB) phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB | Total
Number analyzed (Participants) | 267 | 265 | 266 | 798
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 49 | 49 | 47 | 145
  Between 18 and 65 years | 210 | 206 | 207 | 623
  >=65 years | 8 | 10 | 12 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 117 | 116 | 359
  Male | 141 | 148 | 150 | 439
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 65 | 62 | 52 | 179
  Not Hispanic or Latino | 200 | 203 | 214 | 617
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 1 | 7
  Asian | 38 | 41 | 45 | 124
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 9 | 10 | 33
  White | 209 | 208 | 204 | 621
  More than one race | 2 | 3 | 5 | 10
  Unknown or Not Reported | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Loss of Response: Double-blind (DB) Period
Description: Percentage of participants with loss of response requiring rescue treatment during double blind period was determined. Loss of response denoted as flare and was define as a loss of at least 50% of EASI total score at Week 12 and with an IGA score of 2 or higher. EASI quantifies severity of participant's atopic dermatitis (AD) based on both severity of lesion clinical signs and % of body surface area (BSA) affected. EASI is a composite scoring by AD clinical evaluator of degree of erythema, induration/papulation, excoriation, and lichenification for each of 4 body regions. EASI total score range from 0.0 to 72.0, with higher scores representing greater severity of AD. IGA assesses severity of AD on 5-point scale (0 to 4, higher scores = more severity), reflecting global consideration of erythema, induration and scaling. Where, 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate and 4 = severe.
Time Frame: From Day 1 of up to Week 40 of double blind period
Population: Full analysis set-randomized (FAS-RA) included as all participants who were randomized at Week 12 and received at least 1 dose of study medication within DB phase. Missing event times were considered as right censored (CAR) on last date of randomized treatment.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 267 | 265 | 266
percentage of participants | 77.5 | 39.6 | 16.5

2. Secondary Outcome: Time to First Loss of Response Based on Investigator's Global Assessment (IGA) Score of 2 or Higher: Double-blind Period
Description: Time (in days) to loss of response based on achieving IGA >=2 (for the first time) as measured from date of first dose of randomized treatment until the last dose of randomized treatment (if not entered rescue) or first day of rescue treatment (if entered rescue). IGA assesses severity of AD on a 5-point scale (0 to 4, higher scores indicated more severity), reflecting global consideration of erythema, induration and scaling. Where, 0 = clear, AD is cleared; 1 = almost clear, AD not entirely cleared, light pink residual lesions; 2 = mild, AD with light red lesions; 3 = moderate, AD with red lesions; 4 = severe, AD with deep, dark red lesions.
Time Frame: From date of first dose of randomized treatment until the last dose of randomized treatment (if not entered rescue) or first day of rescue treatment (if entered rescue) (maximum up to Week 40, visit window +/- 7 Days)
Population: FAS-RA included as all participants who were randomized at Week 12 and received at least one dose of study medication within the double-blind phase. Missing event times were considered as right censored (CAR) on last date of randomized treatment. Here, Overall 'Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 247 | 183 | 145
days | 27.0 (26.0) [26.0 to 28.0] | 78.0 (32.0) [32.0 to 112.0] | 201.0 (177.0) [177.0 to 282.0]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; A Cox regression model with treatment, age group and disease severity as stratification covariates was used to estimate the hazard ratio and the corresponding 95% CI; Test type: Superiority; p < 0.0001, Log Rank — A stratified log-rank test with age group and disease severity as stratification variables was performed to evaluate P value; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.286 to 0.424]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.22, 95% CI 2-sided [0.176 to 0.270]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.503 to 0.780]

3. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) Response of Clear (0) or Almost Clear (1) and a Reduction of Greater Than or Equal to (>=) 2 Points From Baseline at Weeks 12, 16, 28, 40, and 52: Double-blind Period
Description: IGA assessed severity of AD on a 5-point scale (0 to 4, higher scores indicated more severity), reflecting global consideration of erythema, induration and scaling. Where, 0 = clear, AD is cleared; 1 = almost clear, AD not entirely cleared, light pink residual lesions; 2 = mild, AD with light red lesions; 3 = moderate, AD with red lesions; 4 = severe, AD with deep dark red lesions.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: FAS-RA included as all participants who were randomized at Week 12 and received at least 1 dose of study medication within DB phase. Here 'Overall Number of Participants Analyzed' signifies number participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for the specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 267 | 264 | 266
percentage of participants
  Week 12: number analyzed (Participants) | 266 | 264 | 265
  Week 12 | 99.6 [98.9 to 100.0] | 99.6 [98.9 to 100.0] | 99.2 [98.2 to 100.0]
  Week 16: number analyzed (Participants) | 267 | 263 | 266
  Week 16 | 15.4 [11.0 to 19.7] | 55.5 [49.5 to 61.5] | 77.8 [72.8 to 82.8]
  Week 28: number analyzed (Participants) | 267 | 260 | 262
  Week 28 | 10.5 [6.8 to 14.2] | 45.0 [39.0 to 51.0] | 61.8 [55.9 to 67.7]
  Week 40: number analyzed (Participants) | 265 | 260 | 259
  Week 40 | 10.6 [6.9 to 14.3] | 42.3 [36.3 to 48.3] | 57.1 [51.1 to 63.2]
  Week 52: number analyzed (Participants) | 264 | 258 | 257
  Week 52 | 11.7 [7.9 to 15.6] | 36.8 [30.9 to 42.7] | 54.1 [48.0 to 60.2]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Week 12: Difference in percentage (PF-04965842 - Placebo) and CI for difference were calculated based on the weighted average of difference for each randomization stratum and disease severity at baseline using the normal approximation of binomial proportions; Test type: Superiority; p = 0.9495, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 0.0, 95% CI 2-sided [-1.0 to 1.1]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.5717, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = -0.4, 95% CI 2-sided [-1.6 to 0.9]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; Week 12: Difference in percentage and CI for difference were calculated based on the weighted average of difference for each randomization stratum and disease severity at baseline using the normal approximation of binomial proportions; Test type: Superiority; Difference in percentage = -0.4, 95% CI 2-sided [-1.7 to 0.9]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Week 16: Difference in percentage (PF-04965842 - Placebo) and CI for difference were calculated based on the weighted average of difference for each randomization stratum and disease severity at baseline using the normal approximation of binomial proportions; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 40.5, 95% CI 2-sided [33.1 to 47.8]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 62.6, 95% CI 2-sided [56.1 to 69.2]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; Week 16: Difference in percentage and CI for difference were calculated based on the weighted average of difference for each randomization stratum and disease severity at baseline using the normal approximation of binomial proportions; Test type: Superiority; Difference in percentage = 22.1, 95% CI 2-sided [14.3 to 29.9]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Week 28: Difference in percentage (PF-04965842 - Placebo) and CI for difference were calculated based on the weighted average of difference for each randomization stratum and disease severity at baseline using the normal approximation of binomial proportions; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 35.1, 95% CI 2-sided [28.1 to 42.0]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 51.5, 95% CI 2-sided [44.6 to 58.4]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; Week 28: Difference in percentage and CI for difference were calculated based on the weighted average of difference for each randomization stratum and disease severity at baseline using the normal approximation of binomial proportions; Test type: Superiority; Difference in percentage = 16.5, 95% CI 2-sided [8.1 to 24.8]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Week 40: Difference in percentage (PF-04965842 - Placebo) and CI for difference were calculated based on the weighted average of difference for each randomization stratum and disease severity at baseline using the normal approximation of binomial proportions; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 32.2, 95% CI 2-sided [25.2 to 39.2]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 46.9, 95% CI 2-sided [39.9 to 53.8]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; Week 40: Difference in percentage and CI for difference were calculated based on the weighted average of difference for each randomization stratum and disease severity at baseline using the normal approximation of binomial proportions; Test type: Superiority; Difference in percentage = 14.2, 95% CI 2-sided [5.9 to 22.6]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Week 52: Difference in percentage (PF-04965842 - Placebo) and CI for difference were calculated based on the weighted average of difference for each randomization stratum and disease severity at baseline using the normal approximation of binomial proportions; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 25.5, 95% CI 2-sided [18.5 to 32.5]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 42.5, 95% CI 2-sided [35.3 to 49.7]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; Week 52: Difference in percentage and CI for difference were calculated based on the weighted average of difference for each randomization stratum and disease severity at baseline using the normal approximation of binomial proportions; Test type: Superiority; Difference in percentage = 17.1, 95% CI 2-sided [8.6 to 25.5]

4. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index (EASI) Response >=50% Improvement From Baseline at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: EASI quantifies severity of participant's AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of BSA affected. Severity of clinical signs of AD (erythema [E], induration/papulation [I], excoriation [Ex] and lichenification [L]) was scored separately for each of 4 body regions (head and neck [h], upper limbs [u], trunk [t] [including axillae and groin] and lower limbs [l] [including buttocks]) on 4-point scale: 0 = absent; 1 = mild; 2 = moderate; 3 = severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score = 0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); where A = area score. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: FAS-RA included as all participants who were randomized at Week 12 and received at least 1 dose of study medication within DB phase. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 267 | 264 | 266
percentage of participants
  Week 12: number analyzed (Participants) | 266 | 264 | 265
  Week 12 | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0]
  Week 16: number analyzed (Participants) | 267 | 263 | 266
  Week 16 | 40.8 [34.9 to 46.7] | 83.3 [78.8 to 87.8] | 96.2 [94.0 to 98.5]
  Week 28: number analyzed (Participants) | 267 | 260 | 262
  Week 28 | 22.8 [17.8 to 27.9] | 68.1 [62.4 to 73.7] | 85.9 [81.7 to 90.1]
  Week 40: number analyzed (Participants) | 265 | 260 | 259
  Week 40 | 16.6 [12.1 to 21.1] | 57.3 [51.3 to 63.3] | 74.9 [69.6 to 80.2]
  Week 52: number analyzed (Participants) | 264 | 258 | 257
  Week 52 | 15.9 [11.5 to 20.3] | 50.8 [44.7 to 56.9] | 71.2 [65.7 to 76.7]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Difference in percentage = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; Week 12: Difference in percentage (PF-04965842 - Placebo) and CI for difference were calculated based on the weighted average of difference for each randomization stratum and disease severity at baseline using the normal approximation of binomial proportions. P-value was adjusted by disease severity at baseline and randomization strata; Test type: Superiority; Difference in percentage = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Difference in percentage = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 42.7, 95% CI 2-sided [35.3 to 50.1]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 55.4, 95% CI 2-sided [49.1 to 61.7]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; Difference in percentage = 12.9, 95% CI 2-sided [7.9 to 17.9]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 45.5, 95% CI 2-sided [37.9 to 53.0]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 63.0, 95% CI 2-sided [56.4 to 69.5]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; Difference in percentage = 17.7, 95% CI 2-sided [10.7 to 24.7]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 41.0, 95% CI 2-sided [33.6 to 48.5]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 58.3, 95% CI 2-sided [51.3 to 65.2]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 12]; Test type: Superiority; Difference in percentage = 17.5, 95% CI 2-sided [9.6 to 25.5]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 35.3, 95% CI 2-sided [27.8 to 42.8]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 13]; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 55.3, 95% CI 2-sided [48.3 to 62.4]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; Difference in percentage = 20.3, 95% CI 2-sided [12.1 to 28.5]

5. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index (EASI) Response >=75% Improvement From Baseline at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: EASI quantifies severity of participant's AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of BSA affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0 = absent; 1 = mild; 2 = moderate; 3 = severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score = 0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll). Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 267 | 264 | 266
percentage of participants
  Week 12: number analyzed (Participants) | 266 | 264 | 265
  Week 12 | 99.2 [98.2 to 100.0] | 100.0 [98.6 to 100.0] | 99.6 [98.9 to 100.0]
  Week 16: number analyzed (Participants) | 267 | 263 | 266
  Week 16 | 27.0 [21.6 to 32.3] | 76.0 [70.9 to 81.2] | 92.5 [89.3 to 95.7]
  Week 28: number analyzed (Participants) | 267 | 260 | 262
  Week 28 | 18.0 [13.4 to 22.6] | 60.4 [54.4 to 66.3] | 80.5 [75.7 to 85.3]
  Week 40: number analyzed (Participants) | 265 | 260 | 259
  Week 40 | 15.1 [10.8 to 19.4] | 54.2 [48.2 to 60.3] | 71.8 [66.3 to 77.3]
  Week 52: number analyzed (Participants) | 264 | 258 | 257
  Week 52 | 14.0 [9.8 to 18.2] | 46.5 [40.4 to 52.6] | 65.8 [60.0 to 71.6]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1848, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 0.7, 95% CI 2-sided [-0.3 to 1.7]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.5971, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 0.3, 95% CI 2-sided [-0.9 to 1.6]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; Difference in percentage = -0.4, 95% CI 2-sided [-1.1 to 0.4]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 49.4, 95% CI 2-sided [42.0 to 56.8]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 65.5, 95% CI 2-sided [59.3 to 71.7]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; Difference in percentage = 16.3, 95% CI 2-sided [10.3 to 22.3]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 42.7, 95% CI 2-sided [35.2 to 50.2]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 62.6, 95% CI 2-sided [56.0 to 69.2]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; Difference in percentage = 19.8, 95% CI 2-sided [12.3 to 27.4]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 39.5, 95% CI 2-sided [32.1 to 46.9]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 56.7, 95% CI 2-sided [49.8 to 63.7]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 12]; Test type: Superiority; Difference in percentage = 17.4, 95% CI 2-sided [9.3 to 25.5]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 33.0, 95% CI 2-sided [25.7 to 40.4]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 51.7, 95% CI 2-sided [44.6 to 58.8]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; Difference in percentage = 19.2, 95% CI 2-sided [10.8 to 27.6]

6. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index (EASI) Response >=90% Improvement From Baseline at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: EASI quantifies severity of participant's AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of BSA affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0 = absent; 1 = mild; 2 = moderate; 3 = severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score = 0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll). Total EASI score ranged from 0.0 to 72.0, higher scores=greater severity of AD.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 267 | 264 | 266
percentage of participants
  Week 12: number analyzed (Participants) | 266 | 264 | 265
  Week 12 | 84.6 [80.2 to 88.9] | 87.1 [83.1 to 91.2] | 86.4 [82.3 to 90.5]
  Week 16: number analyzed (Participants) | 267 | 263 | 266
  Week 16 | 13.9 [9.7 to 18.0] | 51.3 [45.3 to 57.4] | 77.1 [72.0 to 82.1]
  Week 28: number analyzed (Participants) | 267 | 260 | 262
  Week 28 | 10.5 [6.8 to 14.2] | 46.9 [40.9 to 53.0] | 64.5 [58.7 to 70.3]
  Week 40: number analyzed (Participants) | 265 | 260 | 259
  Week 40 | 12.1 [8.2 to 16.0] | 41.5 [35.5 to 47.5] | 58.7 [52.7 to 64.7]
  Week 52: number analyzed (Participants) | 264 | 258 | 257
  Week 52 | 10.6 [6.9 to 14.3] | 37.6 [31.7 to 43.5] | 54.5 [48.4 to 60.6]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.3994, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 2.6, 95% CI 2-sided [-3.3 to 8.4]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.5542, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 1.8, 95% CI 2-sided [-4.1 to 7.8]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; Difference in percentage = -0.8, 95% CI 2-sided [-6.5 to 5.0]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 37.5, 95% CI 2-sided [30.2 to 44.9]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 63.3, 95% CI 2-sided [56.8 to 69.8]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; Difference in percentage = 25.5, 95% CI 2-sided [17.7 to 33.4]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 36.9, 95% CI 2-sided [29.9 to 44.0]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 54.2, 95% CI 2-sided [47.3 to 61.0]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; Difference in percentage = 17.2, 95% CI 2-sided [8.9 to 25.5]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 29.8, 95% CI 2-sided [22.7 to 37.0]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 46.7, 95% CI 2-sided [39.6 to 53.8]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 12]; Test type: Superiority; Difference in percentage = 16.9, 95% CI 2-sided [8.5 to 25.3]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 27.4, 95% CI 2-sided [20.4 to 34.3]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 43.8, 95% CI 2-sided [36.7 to 50.9]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; Difference in percentage = 16.8, 95% CI 2-sided [8.4 to 25.2]

7. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index (EASI) Response >=100% Improvement From Baseline at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: EASI quantifies severity of participant's AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of BSA affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll). Total EASI score ranged from 0.0 to 72.0, higher scores=greater severity of AD.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 267 | 264 | 266
percentage of participants
  Week 12: number analyzed (Participants) | 266 | 264 | 265
  Week 12 | 30.5 [24.9 to 36.0] | 30.3 [24.8 to 35.8] | 28.3 [22.9 to 33.7]
  Week 16: number analyzed (Participants) | 267 | 263 | 266
  Week 16 | 3.7 [1.5 to 6.0] | 15.2 [10.9 to 19.5] | 28.9 [23.5 to 34.4]
  Week 28: number analyzed (Participants) | 267 | 260 | 262
  Week 28 | 4.1 [1.7 to 6.5] | 16.5 [12.0 to 21.1] | 30.2 [24.6 to 35.7]
  Week 40: number analyzed (Participants) | 265 | 260 | 259
  Week 40 | 4.5 [2.0 to 7.0] | 15.8 [11.3 to 20.2] | 30.1 [24.5 to 35.7]
  Week 52: number analyzed (Participants) | 264 | 258 | 257
  Week 52 | 4.5 [2.0 to 7.1] | 18.6 [13.9 to 23.4] | 28.8 [23.3 to 34.3]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.9313, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 0.3, 95% CI 2-sided [-7.5 to 8.1]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.6043, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = -2.1, 95% CI 2-sided [-9.8 to 5.7]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; Difference in percentage = -2.3, 95% CI 2-sided [-10.0 to 5.4]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 11.6, 95% CI 2-sided [6.6 to 16.5]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 25.3, 95% CI 2-sided [19.4 to 31.2]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; Difference in percentage = 13.5, 95% CI 2-sided [6.6 to 20.4]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 12.9, 95% CI 2-sided [7.7 to 18.0]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 26.0, 95% CI 2-sided [19.9 to 32.0]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; Difference in percentage = 13.4, 95% CI 2-sided [6.3 to 20.6]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 11.7, 95% CI 2-sided [6.5 to 16.8]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 25.7, 95% CI 2-sided [19.6 to 31.8]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 12]; Test type: Superiority; Difference in percentage = 14.1, 95% CI 2-sided [7.0 to 21.2]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 14.6, 95% CI 2-sided [9.2 to 20.0]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 24.5, 95% CI 2-sided [18.4 to 30.5]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; Difference in percentage = 10.0, 95% CI 2-sided [2.7 to 17.2]

8. Secondary Outcome: Percentage of Participants With Greater Than or Equal 4 Points Improvement in the Numerical Rating Scale (NRS) for Severity of Pruritus From Baseline at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: Participants were asked to assess their worst itching due to AD over the past 24 hours on an NRS scale ranged from 0 (no itch) to 10 (worst itch imaginable), where higher scores indicated worse disease status.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 258 | 254 | 250
percentage of participants
  Week 12: number analyzed (Participants) | 230 | 237 | 232
  Week 12 | 82.2 [77.2 to 87.1] | 84.0 [79.3 to 88.6] | 81.9 [76.9 to 86.9]
  Week 16: number analyzed (Participants) | 252 | 251 | 250
  Week 16 | 15.9 [11.4 to 20.4] | 54.6 [48.4 to 60.7] | 75.6 [70.3 to 80.9]
  Week 28: number analyzed (Participants) | 258 | 251 | 245
  Week 28 | 11.6 [7.7 to 15.5] | 45.0 [38.9 to 51.2] | 66.9 [61.0 to 72.8]
  Week 40: number analyzed (Participants) | 257 | 254 | 246
  Week 40 | 10.1 [6.4 to 13.8] | 39.4 [33.4 to 45.4] | 55.7 [49.5 to 61.9]
  Week 52: number analyzed (Participants) | 252 | 217 | 204
  Week 52 | 8.3 [4.9 to 11.7] | 27.6 [21.7 to 33.6] | 49.0 [42.2 to 55.9]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.6082, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 1.8, 95% CI 2-sided [-5.0 to 8.5]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.9640, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 0.2, 95% CI 2-sided [-6.7 to 7.0]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; Difference in percentage = -2.4, 95% CI 2-sided [-9.1 to 4.4]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 38.9, 95% CI 2-sided [31.2 to 46.5]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 59.7, 95% CI 2-sided [52.7 to 66.7]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; Difference in percentage = 20.9, 95% CI 2-sided [12.7 to 29.0]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 33.9, 95% CI 2-sided [26.6 to 41.2]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 55.3, 95% CI 2-sided [48.2 to 62.3]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; Difference in percentage = 21.7, 95% CI 2-sided [13.2 to 30.2]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 29.7, 95% CI 2-sided [22.7 to 36.7]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 45.5, 95% CI 2-sided [38.4 to 52.7]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 12]; Test type: Superiority; Difference in percentage = 16.0, 95% CI 2-sided [7.4 to 24.6]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 19.9, 95% CI 2-sided [13.0 to 26.8]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 40.5, 95% CI 2-sided [32.8 to 48.1]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; Difference in percentage = 20.9, 95% CI 2-sided [11.8 to 30.0]

9. Secondary Outcome: Percent Change From Baseline in Body Surface Area (BSA) at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: 4 body regions evaluated: head and neck, upper limbs, trunk (including axillae, groin/genitals), lower limbs (including buttocks) excluding scalp, palms, soles. BSA calculated by handprint method. Number (No) of handprints (size of participant's hand with fingers in closed position) fitting in affected area of a body region was estimated. Maximum No of handprints were 10, 20, 30, 40 for head and neck, upper limbs, trunk, and lower limbs respectively. Surface area (SA) of body region equivalent to 1 handprint: 1 handprint=10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. %Change BSA for a body region was calculated as=total No of handprints in a body region* %SA equivalent to 1 handprint. %BSA for an individual: arithmetic mean of %BSA of all 4 body regions, ranged from 0-100%, higher values=greater AD severity.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 266 | 264 | 265
percent change
  Change at Week 12 | -95.6 [-100.0 to -88.5] | -96.7 [-100.0 to -91.5] | -96.7 [-100.0 to -89.2]
  Change at Week 16: number analyzed (Participants) | 135 | 223 | 256
  Change at Week 16 | -68.5 [-89.8 to -37.5] | -90.9 [-97.6 to -78.3] | -96.3 [-100.0 to -88.7]
  Change at Week 28: number analyzed (Participants) | 64 | 180 | 227
  Change at Week 28 | -85.2 [-95.8 to -63.5] | -93.8 [-99.5 to -81.4] | -96.4 [-100.0 to -85.7]
  Change at Week 40: number analyzed (Participants) | 46 | 151 | 197
  Change at Week 40 | -91.2 [-100.0 to -77.9] | -95.8 [-100.0 to -83.5] | -96.8 [-100.0 to -88.8]
  Change at Week 52: number analyzed (Participants) | 42 | 134 | 185
  Change at Week 52 | -91.5 [-100.0 to -77.9] | -96.9 [-100.0 to -83.4] | -96.9 [-100.0 to -88.2]

10. Secondary Outcome: Percent Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Total Score at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: SCORAD: scoring index for AD combining extent (A), severity (B), subjective symptoms (C). A: rule of 9 used to calculate BSA affected by AD as % of whole BSA for each body region- head and neck 9%; upper limbs 9% each; lower limbs 18% each; anterior trunk 18%; back 18%; genitals 1%. Score of each body region added to determine A (0-100). B: severity of each sign (erythema; edema; oozing; excoriation; skin thickening; dryness) was assessed as none (0), mild (1), moderate (2), severe (3); severity scores added to give B (0-18). C: pruritus and sleep loss, each of these 2 were scored by participant/caregiver using VAS where, 0=no itch/no sleep loss and 10=worst imaginable itch/sleep loss, higher scores=worse symptoms. Scores for itch and sleep loss added to give 'C' (0-20). SCORAD calculated as: A/5+7*B/2+C; range (0-103); higher values=worse outcome.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 265 | 264 | 265
percent change
  Change at Week 12 | -84.0 [-94.7 to -73.5] | -84.4 [-95.2 to -74.9] | -84.4 [-93.8 to -74.2]
  Change at Week 16: number analyzed (Participants) | 134 | 224 | 256
  Change at Week 16 | -50.4 [-68.3 to -32.1] | -71.7 [-87.8 to -60.5] | -83.6 [-95.1 to -70.6]
  Change at Week 28: number analyzed (Participants) | 62 | 177 | 227
  Change at Week 28 | -63.4 [-81.9 to -48.3] | -77.8 [-90.2 to -62.6] | -83.8 [-97.4 to -66.4]
  Change at Week 40: number analyzed (Participants) | 46 | 152 | 196
  Change at Week 40 | -74.4 [-89.5 to -60.6] | -77.1 [-94.1 to -64.3] | -84.6 [-98.6 to -68.4]
  Change at Week 52: number analyzed (Participants) | 43 | 132 | 184
  Change at Week 52 | -73.3 [-89.8 to -58.0] | -82.5 [-97.7 to -64.1] | -83.2 [-100.0 to -69.1]

11. Secondary Outcome: Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Visual Analogue Scale (VAS) of Itch and Sleep Loss at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: SCORAD: scoring index for AD combining extent (A), severity (B), subjective symptoms (C). A: rule of 9 used to calculate BSA affected by AD as % of whole BSA for each body region-head and neck 9%; upper limbs 9% each; lower limbs 18% each; anterior trunk 18%; back 18%; genitals 1%. Score of each body region added to determine A (0-100). B: severity of each sign (erythema; edema; oozing; excoriation; skin thickening; dryness) was assessed as none (0), mild (1), moderate (2), severe (3). Severity scores added to give B (0-18). C: pruritus and sleep loss, each were scored by participant/caregiver using VAS where, 0=no itch/no sleep loss and 10=worst imaginable itch/sleep loss, higher scores=worse symptoms. Scores for itch and sleep loss added to give 'C' (0-20). SCORAD calculated as: A/5+7*B/2+C; range (0-103); higher values=worse outcome.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 264 | 264 | 261
units on a scale
  Pruritus VAS: Change at Week 12 | -6.1 [-6.3 to -5.9] | -6.1 [-6.3 to -5.9] | -6.1 [-6.3 to -5.9]
  Pruritus VAS: Change at Week 16 | 3.4 [3.0 to 3.7] | 1.2 [1.0 to 1.5] | 0.2 [-0.1 to 0.4]
  Pruritus VAS: Change at Week 28 | 2.4 [1.9 to 2.9] | 1.1 [0.8 to 1.4] | 0.5 [0.3 to 0.8]
  Pruritus VAS: Change at Week 40 | 2.2 [1.6 to 2.8] | 1.2 [0.9 to 1.6] | 0.4 [0.1 to 0.7]
  Pruritus VAS: Change at Week 52 | 1.8 [1.2 to 2.4] | 1.3 [0.9 to 1.6] | 0.5 [0.2 to 0.8]
  Sleep Loss VAS: Change at Week 12: number analyzed (Participants) | 264 | 264 | 260
  Sleep Loss VAS: Change at Week 12 | -5.0 [-5.2 to -4.8] | -5.0 [-5.2 to -4.8] | -5.1 [-5.3 to -4.9]
  Sleep Loss VAS: Change at Week 16: number analyzed (Participants) | 264 | 264 | 260
  Sleep Loss VAS: Change at Week 16 | 2.3 [2.0 to 2.6] | 0.5 [0.3 to 0.8] | 0.0 [-0.2 to 0.2]
  Sleep Loss VAS: Change at Week 28: number analyzed (Participants) | 264 | 264 | 260
  Sleep Loss VAS: Change at Week 28 | 1.3 [0.9 to 1.7] | 0.6 [0.4 to 0.9] | 0.2 [0.0 to 0.4]
  Sleep Loss VAS: Change at Week 40: number analyzed (Participants) | 264 | 264 | 260
  Sleep Loss VAS: Change at Week 40 | 1.3 [0.8 to 1.8] | 0.6 [0.3 to 0.9] | 0.2 [0.0 to 0.4]
  Sleep Loss VAS: Change at Week 52: number analyzed (Participants) | 264 | 264 | 260
  Sleep Loss VAS: Change at Week 52 | 1.2 [0.7 to 1.8] | 0.9 [0.5 to 1.2] | 0.3 [0.0 to 0.5]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Pruritus VAS: Week 12: The least squares mean (LSM) differences between treatment groups were derived from the statistical model. Mixed model repeated measure (MMRM) contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p = 0.9207, Mixed Models Analysis; LSM difference = 0.0, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; Pruritus VAS: Week 12: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p = 0.9998, Mixed Models Analysis; LSM difference = 0.0, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; LSM difference = 0.0, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Pruritus VAS: Week 16: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -2.1, 95% CI 2-sided [-2.5 to -1.7]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -3.2, 95% CI 2-sided [-3.6 to -2.8]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; LSM difference = -1.1, 95% CI 2-sided [-1.4 to -0.7]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Pruritus VAS: Week 28: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.4, 95% CI 2-sided [-2.0 to -0.8]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.9, 95% CI 2-sided [-2.5 to -1.3]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; LSM difference = -0.5, 95% CI 2-sided [-0.9 to -0.1]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Pruritus VAS: Week 40: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p = 0.0039, Mixed Models Analysis; LSM difference = -1.0, 95% CI 2-sided [-1.7 to -0.3]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.8, 95% CI 2-sided [-2.5 to -1.2]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; LSM difference = -0.8, 95% CI 2-sided [-1.3 to -0.4]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Pruritus VAS: Week 52: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p = 0.1488, Mixed Models Analysis; LSM difference = -0.5, 95% CI 2-sided [-1.2 to 0.2]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 13]; Test type: Superiority; p = 0.0003, Mixed Models Analysis; LSM difference = -1.3, 95% CI 2-sided [-2.0 to -0.6]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 13]; Test type: Superiority; LSM difference = -0.8, 95% CI 2-sided [-1.2 to -0.3]
Statistical Analysis 16: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Sleep Loss VAS: Week 12: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p = 0.9294, Mixed Models Analysis; LSM difference = 0.0, 95% CI 2-sided [-0.2 to 0.2]
Statistical Analysis 17: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 16]; Test type: Superiority; p = 0.4081, Mixed Models Analysis; LSM difference = -0.1, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 18: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 16]; Test type: Superiority; LSM difference = -0.1, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 19: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Sleep Loss VAS: Week 16: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.8, 95% CI 2-sided [-2.1 to -1.4]
Statistical Analysis 20: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 19]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -2.3, 95% CI 2-sided [-2.7 to -2.0]
Statistical Analysis 21: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 19]; Test type: Superiority; LSM difference = -0.6, 95% CI 2-sided [-0.9 to -0.2]
Statistical Analysis 22: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Sleep Loss VAS: Week 28: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p = 0.0035, Mixed Models Analysis; LSM difference = -0.7, 95% CI 2-sided [-1.2 to -0.2]
Statistical Analysis 23: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 22]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.2, 95% CI 2-sided [-1.6 to -0.7]
Statistical Analysis 24: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 22]; Test type: Superiority; LSM difference = -0.5, 95% CI 2-sided [-0.8 to -0.1]
Statistical Analysis 25: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Sleep Loss VAS: Week 40: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p = 0.0136, Mixed Models Analysis; LSM difference = -0.7, 95% CI 2-sided [-1.2 to -0.1]
Statistical Analysis 26: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 25]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.1, 95% CI 2-sided [-1.6 to -0.6]
Statistical Analysis 27: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 25]; Test type: Superiority; LSM difference = -0.4, 95% CI 2-sided [-0.8 to 0.0]
Statistical Analysis 28: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Sleep Loss VAS: Week 52: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p = 0.2887, Mixed Models Analysis; LSM difference = -0.3, 95% CI 2-sided [-1.0 to 0.3]
Statistical Analysis 29: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 28]; Test type: Superiority; p = 0.0025, Mixed Models Analysis; LSM difference = -1.0, 95% CI 2-sided [-1.6 to -0.3]
Statistical Analysis 30: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 11, analysis 28]; Test type: Superiority; LSM difference = -0.6, 95% CI 2-sided [-1.0 to -0.2]

12. Secondary Outcome: Percentage of Participants With >=50% Improvement From Baseline in Scoring Atopic Dermatitis (SCORAD) Response at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: SCORAD: scoring index for AD combining extent (A), severity (B), subjective symptoms (C). A: rule of 9 used to calculate BSA affected by AD as % of whole BSA for each body region- head and neck 9%; upper limbs 9% each; lower limbs 18% each; anterior trunk 18%; back 18%; genitals 1%. Score of each body region added to determine A (0-100). B: severity of each sign (erythema; edema; oozing; excoriation; skin thickening; dryness) was assessed as none (0), mild (1), moderate (2), severe (3). Severity scores added to give B (0-18). C: pruritus and sleep loss, each were scored by participant/caregiver using VAS where, 0=no itch/no sleep loss and 10=worst imaginable itch/sleep loss, higher scores=worse symptoms. Scores for itch and sleep loss added to give 'C' (0-20). SCORAD calculated as: A/5+7*B/2+C; range (0-103); higher values=worse outcome.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 266 | 264 | 266
percentage of participants
  Week 12: number analyzed (Participants) | 265 | 264 | 265
  Week 12 | 97.4 [95.4 to 99.3] | 98.5 [97.0 to 100.0] | 97.0 [94.9 to 99.0]
  Week 16 | 25.6 [20.3 to 30.8] | 72.0 [66.6 to 77.4] | 89.1 [85.4 to 92.8]
  Week 28: number analyzed (Participants) | 266 | 259 | 263
  Week 28 | 15.8 [11.4 to 20.2] | 56.8 [50.7 to 62.8] | 75.7 [70.5 to 80.9]
  Week 40: number analyzed (Participants) | 264 | 260 | 258
  Week 40 | 14.4 [10.2 to 18.6] | 51.2 [45.1 to 57.2] | 69.0 [63.3 to 74.6]
  Week 52: number analyzed (Participants) | 264 | 258 | 257
  Week 52 | 14.8 [10.5 to 19.1] | 44.6 [38.5 to 50.6] | 65.8 [60.0 to 71.6]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4244, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 1.0, 95% CI 2-sided [-1.4 to 3.4]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.8092, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = -0.3, 95% CI 2-sided [-3.1 to 2.4]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; Difference in percentage = -1.5, 95% CI 2-sided [-4.1 to 1.0]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 46.7, 95% CI 2-sided [39.2 to 54.2]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 63.6, 95% CI 2-sided [57.2 to 70.0]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; Difference in percentage = 17.0, 95% CI 2-sided [10.4 to 23.5]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 41.3, 95% CI 2-sided [33.9 to 48.7]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 59.9, 95% CI 2-sided [53.1 to 66.7]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; Difference in percentage = 18.7, 95% CI 2-sided [10.8 to 26.6]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 37.0, 95% CI 2-sided [29.6 to 44.4]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 54.6, 95% CI 2-sided [47.6 to 61.7]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 12]; Test type: Superiority; Difference in percentage = 17.7, 95% CI 2-sided [9.4 to 26.0]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 30.0, 95% CI 2-sided [22.6 to 37.4]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 50.9, 95% CI 2-sided [43.8 to 58.1]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; Difference in percentage = 21.1, 95% CI 2-sided [12.8 to 29.5]

13. Secondary Outcome: Percentage of Participants With >=75% Improvement From Baseline in Scoring Atopic Dermatitis (SCORAD) Response at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: as for outcome 12
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 266 | 264 | 266
percentage of participants
  Week 12: number analyzed (Participants) | 265 | 264 | 265
  Week 12 | 73.6 [68.3 to 78.9] | 75.0 [69.8 to 80.2] | 71.3 [65.9 to 76.8]
  Week 16 | 9.4 [5.9 to 12.9] | 38.3 [32.4 to 44.1] | 67.3 [61.7 to 72.9]
  Week 28: number analyzed (Participants) | 266 | 259 | 263
  Week 28 | 7.5 [4.3 to 10.7] | 37.8 [31.9 to 43.7] | 56.3 [50.3 to 62.3]
  Week 40: number analyzed (Participants) | 264 | 260 | 258
  Week 40 | 8.3 [5.0 to 11.7] | 32.7 [27.0 to 38.4] | 47.7 [41.6 to 53.8]
  Week 52: number analyzed (Participants) | 264 | 258 | 257
  Week 52 | 7.6 [4.4 to 10.8] | 31.8 [26.1 to 37.5] | 45.9 [39.8 to 52.0]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.7232, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 1.4, 95% CI 2-sided [-6.1 to 8.8]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.5694, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = -2.2, 95% CI 2-sided [-9.8 to 5.4]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; Difference in percentage = -3.7, 95% CI 2-sided [-11.2 to 3.8]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 29.0, 95% CI 2-sided [22.2 to 35.8]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 57.9, 95% CI 2-sided [51.2 to 64.5]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; Difference in percentage = 28.9, 95% CI 2-sided [20.8 to 37.0]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 30.5, 95% CI 2-sided [23.9 to 37.2]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 48.9, 95% CI 2-sided [42.1 to 55.6]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; Difference in percentage = 18.2, 95% CI 2-sided [9.8 to 26.6]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 25.0, 95% CI 2-sided [18.4 to 31.5]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 39.6, 95% CI 2-sided [32.7 to 46.5]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 12]; Test type: Superiority; Difference in percentage = 14.5, 95% CI 2-sided [6.3 to 22.8]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 24.7, 95% CI 2-sided [18.1 to 31.2]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 38.5, 95% CI 2-sided [31.6 to 45.3]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; Difference in percentage = 13.9, 95% CI 2-sided [5.6 to 22.3]

14. Secondary Outcome: Percentage of Participants Achieving IGA Response of Clear (0) or Almost Clear (1) and Greater Than or Equal to (>=) 2 Points Improvement From Rescue Baseline at Rescue Weeks 2, 4, 8 and 12: Rescue Period
Description: IGA assessed severity of AD on a 5-point scale (0-4, higher scores indicated more severity), reflecting global consideration of erythema, induration and scaling. Where, 0=clear, AD is cleared; 1 = almost clear, AD not entirely cleared, light pink residual lesions; 2 = mild, AD with light red lesions; 3 = moderate, AD with red lesions; 4 = severe, AD with deep, dark red lesions.
Time Frame: Rescue Baseline: last observation collected between last dose of blinded treatment and Day 1 (first dose day) of rescue treatment, Rescue Weeks 2, 4, 8 and 12
Population: Full analysis set-rescue (FAS-RE) included all participants who met the protocol definition of a flare during the DB phase and received at least 1 dose of rescue treatment. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg Rescue Period
Number analyzed (Participants) | 342
percentage of participants
  Rescue Week 2: number analyzed (Participants) | 332
  Rescue Week 2 | 30.7 [25.8 to 35.7]
  Rescue Week 4: number analyzed (Participants) | 337
  Rescue Week 4 | 54.6 [49.3 to 59.9]
  Rescue Week 8 | 60.2 [55.0 to 65.4]
  Rescue Week 12: number analyzed (Participants) | 337
  Rescue Week 12 | 64.1 [59.0 to 69.2]

15. Secondary Outcome: Percent Change From Rescue Baseline in Total Eczema Area and Severity Index (EASI) Score at Rescue Weeks 2, 4, 8 and 12: Rescue Period
Description: as for outcome 7
Time Frame: as for outcome 14
Population: FAS-RE included all participants who met the protocol definition of a flare during the DB phase and received at least 1 dose of rescue treatment. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | PF-04965842 200 mg Rescue Period
Number analyzed (Participants) | 348
percent change
  Change at Rescue Week 2 | -71.1 (-73.7) [-73.7 to -68.5]
  Change at Rescue Week 4 | -82.0 (-84.2) [-84.2 to -79.7]
  Change at Rescue Week 8 | -86.4 (-88.2) [-88.2 to -84.6]
  Change at Rescue Week 12 | -87.3 (-89.4) [-89.4 to -85.3]

16. Secondary Outcome: Percentage of Participants Achieving Greater Than or Equal to 4 Points Improvement From Rescue Baseline in Peak Pruritus Numeric Rating Scale (PP-NRS) at Rescue Weeks 2, 4, 8 and 12: Rescue Period
Description: Participants were asked to assess their worst itching due to AD over the past 24 hours on an NRS scale ranged from 0 (no itch) to 10 (worst itch imaginable), where higher scores indicated greater severity.
Time Frame: as for outcome 14
Population: FAS-RE included all participants who met the protocol definition of a flare during the DB phase and received at least 1 dose of rescue treatment. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg Rescue Period
Number analyzed (Participants) | 272
percentage of participants
  Rescue Week 2 | 56.6 [50.7 to 62.5]
  Rescue Week 4: number analyzed (Participants) | 250
  Rescue Week 4 | 63.2 [57.2 to 69.2]
  Rescue Week 8: number analyzed (Participants) | 253
  Rescue Week 8 | 67.2 [61.4 to 73.0]
  Rescue Week 12: number analyzed (Participants) | 153
  Rescue Week 12 | 56.2 [48.3 to 64.1]

17. Secondary Outcome: Percent Change From Rescue Baseline in Percent Body Surface Area (BSA) at Rescue Weeks 2, 4, 8 and 12: Rescue Period
Description: 4 body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin/genitals) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's hand with fingers in a closed position) fitting in affected area of a body region was estimated. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint was equal to 10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Overall % BSA for an individual % BSA of all 4 body regions, ranged from 0 to 100%, with higher values representing greater severity of AD.
Time Frame: as for outcome 14
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | PF-04965842 200 mg Rescue Period
Number analyzed (Participants) | 348
percent change
  Change at Rescue Week 2 | -62.8 [-66.0 to -59.6]
  Change at Rescue Week 4 | -76.4 [-79.1 to -73.7]
  Change at Rescue Week 8 | -82.1 [-84.5 to -79.6]
  Change at Rescue Week 12 | -83.3 [-86.0 to -80.5]

18. Secondary Outcome: Percent Change From Rescue Baseline in Scoring Atopic Dermatitis (SCORAD) Visual Analog Scale (VAS) Score of Itch and Sleep Loss at Rescue Weeks 2, 4, 8 and 12: Rescue Period
Description: as for outcome 12
Time Frame: as for outcome 14
Population: FAS-RE included all participants who met the protocol definition of a flare during the DB phase and received at least 1 dose of rescue treatment.. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | PF-04965842 200 mg Rescue Period
Number analyzed (Participants) | 347
percent change
  Pruritus VAS: Change at Rescue Week 2 | -57.3 (-61.7) [-61.7 to -52.9]
  Pruritus VAS: Change at Rescue Week 4 | -67.5 (-71.3) [-71.3 to -63.7]
  Pruritus VAS: Change at Rescue Week 8 | -68.6 (-73.6) [-73.6 to -63.7]
  Pruritus VAS: Change at Rescue Week 12 | -67.3 (-72.8) [-72.8 to -61.8]
  Sleep Loss VAS: Change at Rescue Week 2 | -62.5 (-69.1) [-69.1 to -55.9]
  Sleep Loss VAS: Change at Rescue Week 4 | -72.4 (-78.6) [-78.6 to -66.3]
  Sleep Loss VAS: Change at Rescue Week 8 | -75.8 (-82.0) [-82.0 to -69.5]
  Sleep Loss VAS: Change at Rescue Week 12 | -74.5 (-81.4) [-81.4 to -67.5]

19. Secondary Outcome: Percentage of Participants With 50% Improvement in Scoring Atopic Dermatitis (SCORAD) From Rescue Baseline at Rescue Weeks 2, 4, 8 and 12: Rescue Period
Description: as for outcome 12
Time Frame: as for outcome 14
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg Rescue Period
Number analyzed (Participants) | 339
percentage of participants
  Rescue Week 2: number analyzed (Participants) | 331
  Rescue Week 2 | 55.0 [49.6 to 60.3]
  Rescue Week 4 | 76.1 [71.6 to 80.6]
  Rescue Week 8: number analyzed (Participants) | 338
  Rescue Week 8 | 79.6 [75.3 to 83.9]
  Rescue Week 12: number analyzed (Participants) | 337
  Rescue Week 12 | 79.8 [75.5 to 84.1]

20. Secondary Outcome: Percentage of Participants With 75% Improvement in Scoring Atopic Dermatitis (SCORAD) From Rescue Baseline at Rescue Weeks 2, 4, 8 and 12: Rescue Period
Description: as for outcome 12
Time Frame: as for outcome 14
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg Rescue Period
Number analyzed (Participants) | 339
percentage of participants
  Rescue Week 2: number analyzed (Participants) | 331
  Rescue Week 2 | 16.9 [12.9 to 21.0]
  Rescue Week 4 | 33.9 [28.9 to 39.0]
  Rescue Week 8: number analyzed (Participants) | 338
  Rescue Week 8 | 44.4 [39.1 to 49.7]
  Rescue Week 12: number analyzed (Participants) | 337
  Rescue Week 12 | 45.4 [40.1 to 50.7]

21. Secondary Outcome: Percentage of Participants Achieving Patient Global Assessment (PtGA) Response of 'Clear (0)' or 'Almost Clear (1)' and Greater Than or Equal to 2 Points Improvement From Baseline at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: Participant responded to the following question: "Overall, how would you describe your Atopic Dermatitis right now?" on a 5-point scale: 0= clear; 1= almost clear; 2= mild; 3= moderate; and 4= severe. Higher scores indicated more severity.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 254 | 262 | 259
percentage of participants
  Week 12: number analyzed (Participants) | 253 | 262 | 258
  Week 12 | 61.7 [55.7 to 67.7] | 64.5 [58.7 to 70.3] | 59.7 [53.7 to 65.7]
  Week 16 | 5.9 [3.0 to 8.8] | 29.8 [24.2 to 35.3] | 48.3 [42.2 to 54.3]
  Week 28: number analyzed (Participants) | 253 | 259 | 256
  Week 28 | 6.3 [3.3 to 9.3] | 30.9 [25.3 to 36.5] | 46.9 [40.8 to 53.0]
  Week 40: number analyzed (Participants) | 252 | 257 | 250
  Week 40 | 7.5 [4.3 to 10.8] | 26.1 [20.7 to 31.4] | 42.0 [35.9 to 48.1]
  Week 52: number analyzed (Participants) | 251 | 256 | 247
  Week 52 | 7.6 [4.3 to 10.8] | 25.8 [20.4 to 31.1] | 39.7 [33.6 to 45.8]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4815, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 3.0, 95% CI 2-sided [-5.3 to 11.3]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.6748, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = -1.8, 95% CI 2-sided [-10.3 to 6.6]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; Difference in percentage = -5.1, 95% CI 2-sided [-13.4 to 3.2]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 24.0, 95% CI 2-sided [17.8 to 30.3]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 42.3, 95% CI 2-sided [35.6 to 49.0]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; Difference in percentage = 18.4, 95% CI 2-sided [10.2 to 26.6]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 24.6, 95% CI 2-sided [18.2 to 31.0]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 40.5, 95% CI 2-sided [33.7 to 47.3]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; Difference in percentage = 15.9, 95% CI 2-sided [7.6 to 24.1]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 18.8, 95% CI 2-sided [12.6 to 25.1]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 34.5, 95% CI 2-sided [27.6 to 41.5]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 12]; Test type: Superiority; Difference in percentage = 15.6, 95% CI 2-sided [7.5 to 23.7]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 18.7, 95% CI 2-sided [12.4 to 25.0]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by disease severity at baseline and randomization strata; Difference in percentage = 32.3, 95% CI 2-sided [25.4 to 39.2]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; Difference in percentage = 13.7, 95% CI 2-sided [5.6 to 21.7]

22. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score for Adults at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: DLQI was a 10-item questionnaire that measures the impact of skin disease. Each question was evaluated on a 4-point scale (range 0 to 3) where, 0 = not at all, 1= a little, 2= a lot, 3= very much, where higher scores indicated more impact on quality of life. Scores from all 10 questions were added up to give DLQI total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: FAS-RA included as all participants who were randomized at Week 12 and received at least 1 dose of study medication within DB phase. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for adults, aged 18 years and above.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 217 | 215 | 217
units on a scale
  Change at Week 12 | -13.5 (-13.9) [-13.9 to -13.0] | -13.4 (-13.8) [-13.8 to -12.9] | -13.5 (-14.0) [-14.0 to -13.1]
  Change at Week 16 | 6.9 (6.1) [6.1 to 7.8] | 1.9 (1.2) [1.2 to 2.5] | 0.4 (-0.2) [-0.2 to 1.0]
  Change at Week 28 | 6.1 (5.0) [5.0 to 7.1] | 2.1 (1.4) [1.4 to 2.7] | 0.9 (0.3) [0.3 to 1.5]
  Change at Week 40 | 4.4 (3.0) [3.0 to 5.7] | 2.5 (1.7) [1.7 to 3.2] | 1.1 (0.5) [0.5 to 1.8]
  Change at Week 52 | 3.6 (2.1) [2.1 to 5.0] | 2.8 (2.0) [2.0 to 3.6] | 0.9 (0.2) [0.2 to 1.6]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Week 12: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p = 0.7373, Mixed Models Analysis; LSM difference = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.8092, Mixed Models Analysis; LSM difference = -0.1, 95% CI 2-sided [-0.7 to 0.5]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; LSM difference = -0.2, 95% CI 2-sided [-0.8 to 0.4]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Week 16: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -5.1, 95% CI 2-sided [-6.1 to -4.0]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -6.6, 95% CI 2-sided [-7.6 to -5.5]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; LSM difference = -1.5, 95% CI 2-sided [-2.4 to -0.6]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Week 28: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -4.0, 95% CI 2-sided [-5.3 to -2.7]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -5.2, 95% CI 2-sided [-6.4 to -3.9]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; LSM difference = -1.2, 95% CI 2-sided [-2.1 to -0.3]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Week 40: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p = 0.0150, Mixed Models Analysis; LSM difference = -1.9, 95% CI 2-sided [-3.5 to -0.4]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -3.2, 95% CI 2-sided [-4.7 to -1.7]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; LSM difference = -1.3, 95% CI 2-sided [-2.3 to -0.3]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; Week 52: The LSM differences between treatment groups were derived from the statistical model. MMRM contained fixed factors of treatment, visit, treatment by visit interaction, baseline disease severity, randomization strata, baseline value and an unstructured covariance matrix; Test type: Superiority; p = 0.3616, Mixed Models Analysis; LSM difference = -0.8, 95% CI 2-sided [-2.4 to 0.9]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; p = 0.0012, Mixed Models Analysis; LSM difference = -2.7, 95% CI 2-sided [-4.3 to -1.1]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; LSM difference = -1.9, 95% CI 2-sided [-3.0 to -0.8]

23. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) Score for Adolescents at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: CDLQI is a 10-item questionnaire that measures the impact of skin disease on adolescents (aged 12-17 years) quality of life over the last week. Each question was evaluated on a 4-point scale (range 0 to 3) where, 0 = not at all , 1 = only a little, 2 = quite a lot, 3 = very much, where higher scores indicated more impact on quality of life. Scores from all 10 questions were added up to give CDLQI total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of children.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: FAS-RA included as all participants who were randomized at Week 12 and received at least 1 dose of study medication within DB phase. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for adolescents, aged 12-17 years.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 49 | 48 | 47
units on a scale
  Change at Week 12 | -9.8 (-10.6) [-10.6 to -8.9] | -9.2 (-10.0) [-10.0 to -8.3] | -9.3 (-10.2) [-10.2 to -8.5]
  Change at Week 16 | 5.9 (4.4) [4.4 to 7.5] | 1.7 (0.5) [0.5 to 2.9] | -0.3 (-1.4) [-1.4 to 0.8]
  Change at Week 28 | 1.5 (-0.2) [-0.2 to 3.2] | 1.6 (0.6) [0.6 to 2.6] | 0.4 (-0.5) [-0.5 to 1.3]
  Change at Week 40 | 2.1 (0.3) [0.3 to 3.8] | 1.7 (0.7) [0.7 to 2.7] | 0.0 (-0.9) [-0.9 to 0.9]
  Change at Week 52 | 2.3 (0.3) [0.3 to 4.4] | 1.3 (0.0) [0.0 to 2.6] | 0.4 (-0.6) [-0.6 to 1.4]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.3339, Mixed Models Analysis; LSM difference = 0.6, 95% CI 2-sided [-0.6 to 1.8]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.4653, Mixed Models Analysis; LSM difference = 0.5, 95% CI 2-sided [-0.8 to 1.7]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; LSM difference = -0.1, 95% CI 2-sided [-1.3 to 1.1]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -4.3, 95% CI 2-sided [-6.2 to -2.3]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -6.2, 95% CI 2-sided [-8.2 to -4.3]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; LSM difference = -2.0, 95% CI 2-sided [-3.6 to -0.3]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p = 0.9083, Mixed Models Analysis; LSM difference = 0.1, 95% CI 2-sided [-1.8 to 2.1]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p = 0.2439, Mixed Models Analysis; LSM difference = -1.1, 95% CI 2-sided [-3.0 to 0.8]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; LSM difference = -1.2, 95% CI 2-sided [-2.6 to 0.1]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; p = 0.7405, Mixed Models Analysis; LSM difference = -0.3, 95% CI 2-sided [-2.4 to 1.7]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; p = 0.0410, Mixed Models Analysis; LSM difference = -2.1, 95% CI 2-sided [-4.1 to -0.1]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; LSM difference = -1.7, 95% CI 2-sided [-3.1 to -0.4]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; p = 0.4026, Mixed Models Analysis; LSM difference = -1.0, 95% CI 2-sided [-3.5 to 1.4]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; p = 0.0944, Mixed Models Analysis; LSM difference = -1.9, 95% CI 2-sided [-4.2 to 0.3]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; LSM difference = -0.9, 95% CI 2-sided [-2.5 to 0.7]

24. Primary Outcome: Time to Loss of Response: Double-blind Period
Description: Time (in days) to loss of response based on achieving IGA >=2 was measured from date of first dose of randomized treatment until last dose of randomized treatment (if not entered rescue) or first day of rescue treatment (if entered rescue) and based on EASI, loss of at least 50% of EASI response at Week 12 and IGA score of 2 or higher. IGA assesses severity of AD on 5-point scale (0 to 4, higher scores=more severity), reflecting global consideration of erythema, induration and scaling with scores 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe. EASI quantifies severity of AD based on severity of lesion clinical signs and % of BSA affected. EASI composite score evaluates degree of erythema, induration/papulation, excoriation, and lichenification.
Time Frame: From date of first dose of randomized treatment until the last dose of randomized treatment (if not entered rescue) or first day of rescue treatment (if entered rescue) (maximum up to Week 40, visit window was extended +/- 45 Days due to COVID 19)
Population: FAS-RA included as all participants who were randomized at Week 12 and received at least 1 dose of study medication within DB phase. Missing event times were considered as right censored (CAR) on last date of randomized treatment. Here 'Overall Number of Participants Analyzed signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 207 | 105 | 44
days | 28.0 [28.0 to 29.0] | 323.0 [282.0 to 323.0] | NA [NA to NA] — Median and 95% CI were not estimable as there were only few participant who had events.
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; A Cox regression model with treatment, age group and disease severity as stratification covariates was used to estimate the hazard ratio and the corresponding 95% confidence interval (CI); Test type: Superiority; p < 0.0001, Log Rank — A stratified log-rank test with age group and disease severity as stratification variables was performed to evaluate p-value; Hazard Ratio (HR) = 0.27, 95% CI 2-sided [0.211 to 0.341]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.10, 95% CI 2-sided [0.070 to 0.136]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.255 to 0.516]

25. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) - Anxiety Scale at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: HADS: participant rated 14-item questionnaire. HADS consisted of 2 subscales: HADS-Anxiety (HADS-A) scale and HADS-Depression (HADS-D) scale, both of these subscales comprised of 7 items each. Each item was rated on a 4-point scale, score range from 0 to 3, where higher scores indicates more anxiety/depression symptoms. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks). HADS-A: sum of all 7 items resulted in score range of 0 (no presence of anxiety) to 21 (severe feeling of anxiety); higher score indicating greater severity of anxiety.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: FAS-RA included as all participants who were randomized at Week 12 and received at least 1 dose of study medication within DB phase. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 266 | 263 | 264
units on a scale
  Change at Week 12 | -2.7 (-3.0) [-3.0 to -2.3] | -2.6 (-2.9) [-2.9 to -2.3] | -2.6 (-2.9) [-2.9 to -2.3]
  Change at Week 16 | 1.4 (1.0) [1.0 to 1.8] | 0.3 (0.0) [0.0 to 0.6] | 0.0 (-0.3) [-0.3 to 0.3]
  Change at Week 28 | 1.0 (0.5) [0.5 to 1.5] | 0.4 (0.1) [0.1 to 0.7] | 0.1 (-0.2) [-0.2 to 0.4]
  Change at Week 40 | 1.0 (0.4) [0.4 to 1.6] | 0.4 (0.1) [0.1 to 0.8] | 0.1 (-0.3) [-0.3 to 0.4]
  Change at Week 52 | 0.8 (0.2) [0.2 to 1.4] | 0.4 (0.1) [0.1 to 0.8] | 0.2 (-0.1) [-0.1 to 0.5]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.7556, Mixed Models Analysis; LSM difference = 0.1, 95% CI 2-sided [-0.4 to 0.6]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.7484, Mixed Models Analysis; LSM difference = 0.1, 95% CI 2-sided [-0.4 to 0.6]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; LSM difference = 0.0, 95% CI 2-sided [-0.5 to 0.5]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.1, 95% CI 2-sided [-1.6 to -0.6]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.4, 95% CI 2-sided [-1.9 to -0.9]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; LSM difference = -0.3, 95% CI 2-sided [-0.7 to 0.1]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p = 0.0242, Mixed Models Analysis; LSM difference = -0.6, 95% CI 2-sided [-1.2 to -0.1]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p = 0.0012, Mixed Models Analysis; LSM difference = -0.9, 95% CI 2-sided [-1.4 to -0.4]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; LSM difference = -0.3, 95% CI 2-sided [-0.6 to 0.1]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; p = 0.1240, Mixed Models Analysis; LSM difference = -0.6, 95% CI 2-sided [-1.3 to 0.2]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; p = 0.0107, Mixed Models Analysis; LSM difference = -0.9, 95% CI 2-sided [-1.6 to -0.2]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; LSM difference = -0.3, 95% CI 2-sided [-0.8 to 0.1]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; p = 0.3139, Mixed Models Analysis; LSM difference = -0.4, 95% CI 2-sided [-1.1 to 0.3]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; p = 0.0853, Mixed Models Analysis; LSM difference = -0.6, 95% CI 2-sided [-1.3 to 0.1]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; LSM difference = -0.2, 95% CI 2-sided [-0.7 to 0.2]

26. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) - Depression Scale at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: HADS: participant rated 14-item questionnaire. HADS consisted of 2 subscales: HADS-A scale and HADS-D scale, both of these subscales comprised of 7 items each. Each item was rated on a 4-point scale, score range from 0 to 3, where higher scores indicates more anxiety/depression symptoms. HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). HADS-D: sum of all 7 items resulted in score range of 0 (no presence of depression) to 21 (severe feeling of depression); higher score indicating greater severity of depression symptoms.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 266 | 263 | 264
units on a scale
  Change at Week 12 | -2.0 (-2.3) [-2.3 to -1.7] | -1.6 (-1.9) [-1.9 to -1.3] | -1.7 (-2.0) [-2.0 to -1.4]
  Change at Week 16 | 1.4 (1.0) [1.0 to 1.8] | 0.0 (-0.3) [-0.3 to 0.3] | 0.0 (-0.2) [-0.2 to 0.3]
  Change at Week 28 | 0.7 (0.2) [0.2 to 1.1] | 0.3 (0.0) [0.0 to 0.5] | 0.1 (-0.2) [-0.2 to 0.4]
  Change at Week 40 | 0.8 (0.2) [0.2 to 1.4] | -0.1 (-0.4) [-0.4 to 0.3] | 0.2 (-0.1) [-0.1 to 0.5]
  Change at Week 52 | 0.4 (-0.1) [-0.1 to 0.9] | -0.1 (-0.4) [-0.4 to 0.2] | 0.1 (-0.2) [-0.2 to 0.3]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.0674, Mixed Models Analysis; LSM difference = 0.4, 95% CI 2-sided [0.0 to 0.8]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.1437, Mixed Models Analysis; LSM difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; LSM difference = -0.1, 95% CI 2-sided [-0.5 to 0.3]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.4, 95% CI 2-sided [-1.8 to -0.9]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.4, 95% CI 2-sided [-1.8 to -0.9]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; LSM difference = 0.0, 95% CI 2-sided [-0.4 to 0.4]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p = 0.1136, Mixed Models Analysis; LSM difference = -0.4, 95% CI 2-sided [-1.0 to 0.1]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p = 0.0276, Mixed Models Analysis; LSM difference = -0.6, 95% CI 2-sided [-1.1 to -0.1]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; LSM difference = -0.2, 95% CI 2-sided [-0.5 to 0.2]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; p = 0.0108, Mixed Models Analysis; LSM difference = -0.9, 95% CI 2-sided [-1.5 to -0.2]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; p = 0.0677, Mixed Models Analysis; LSM difference = -0.6, 95% CI 2-sided [-1.3 to 0.0]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; LSM difference = 0.3, 95% CI 2-sided [-0.2 to 0.7]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; p = 0.1320, Mixed Models Analysis; LSM difference = -0.5, 95% CI 2-sided [-1.1 to 0.1]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; p = 0.2975, Mixed Models Analysis; LSM difference = -0.3, 95% CI 2-sided [-0.9 to 0.3]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; LSM difference = 0.2, 95% CI 2-sided [-0.2 to 0.6]

27. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) Score at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: POEM was a 7-item participant reported outcome (PRO) measure used to assess the impact of AD (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) over the past week. Each item scored as following: no days = 0, 1-2 days = 1, 3-4 days = 2, 5-6 days = 3 and, every day = 4. The total POEM score ranges from 0 to 28, where higher score indicated greater severity.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 265 | 263 | 263
units on a scale
  Change at Week 12 | -15.4 (-16.0) [-16.0 to -14.8] | -15.8 (-16.4) [-16.4 to -15.2] | -15.4 (-16.0) [-16.0 to -14.8]
  Change at Week 16 | 9.8 (8.9) [8.9 to 10.7] | 3.7 (3.0) [3.0 to 4.4] | 0.6 (-0.1) [-0.1 to 1.2]
  Change at Week 28 | 8.3 (6.9) [6.9 to 9.7] | 3.7 (2.8) [2.8 to 4.6] | 1.6 (0.8) [0.8 to 2.4]
  Change at Week 40 | 7.4 (5.8) [5.8 to 9.1] | 4.8 (3.9) [3.9 to 5.8] | 1.9 (1.1) [1.1 to 2.8]
  Change at Week 52 | 7.3 (5.4) [5.4 to 9.2] | 4.9 (3.8) [3.8 to 6.0] | 2.2 (1.3) [1.3 to 3.2]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.3531, Mixed Models Analysis; LSM difference = -0.4, 95% CI 2-sided [-1.3 to 0.4]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.9282, Mixed Models Analysis; LSM difference = 0.0, 95% CI 2-sided [-0.8 to 0.9]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; LSM difference = 0.4, 95% CI 2-sided [-0.4 to 1.3]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -6.1, 95% CI 2-sided [-7.3 to -5.0]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -9.2, 95% CI 2-sided [-10.3 to -8.1]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; LSM difference = -3.1, 95% CI 2-sided [-4.0 to -2.1]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -4.6, 95% CI 2-sided [-6.2 to -2.9]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -6.7, 95% CI 2-sided [-8.3 to -5.1]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; LSM difference = -2.1, 95% CI 2-sided [-3.3 to -0.9]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; p = 0.0082, Mixed Models Analysis; LSM difference = -2.6, 95% CI 2-sided [-4.5 to -0.7]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -5.5, 95% CI 2-sided [-7.4 to -3.6]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; LSM difference = -2.9, 95% CI 2-sided [-4.2 to -1.6]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; p = 0.0313, Mixed Models Analysis; LSM difference = -2.4, 95% CI 2-sided [-4.5 to -0.2]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -5.1, 95% CI 2-sided [-7.1 to -3.0]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; LSM difference = -2.7, 95% CI 2-sided [-4.1 to -1.3]

28. Secondary Outcome: Change From Baseline in Pruritus and Symptoms Assessment for Atopic Dermatitis (PSAAD) Score at Weeks 12, 16, 28, 40 and 52: Double-blind Period
Description: PSAAD is a daily participant reported symptom electronic diary. Participants rated their symptoms of AD over the past 24 hours, using 11 items (itchy skin, painful skin, dry skin, flaky skin, cracked skin, bumpy skin, red skin, discolored skin [darker or lighter], bleeding from skin, seeping or oozing fluid from skin [other than blood], and skin swelling). Participants had to think about all the areas of their body affected by their skin condition and chose the number that best described their experience for each of the 11 items, from 0 (no symptoms) to 10 (extreme symptoms), higher scores signified worse skin condition. Total PSAAD score = arithmetic mean of 11 items, 0 (no symptoms) to 10 (extreme symptoms), where higher score = worse skin condition.
Time Frame: Baseline, Weeks 12, 16, 28, 40 and 52
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB
Number analyzed (Participants) | 254 | 260 | 254
units on a scale
  Change at Week 12 | -4.1 (-4.3) [-4.3 to -3.9] | -4.2 (-4.4) [-4.4 to -4.0] | -4.2 (-4.4) [-4.4 to -4.0]
  Change at Week 16 | 2.1 (1.9) [1.9 to 2.2] | 0.8 (0.6) [0.6 to 0.9] | 0.1 (-0.1) [-0.1 to 0.3]
  Change at Week 28 | 2.3 (2.0) [2.0 to 2.6] | 1.0 (0.8) [0.8 to 1.2] | 0.1 (-0.1) [-0.1 to 0.3]
  Change at Week 40 | 2.0 (1.7) [1.7 to 2.4] | 1.0 (0.8) [0.8 to 1.3] | 0.3 (0.0) [0.0 to 0.5]
  Change at Week 52 | 1.9 (1.5) [1.5 to 2.3] | 1.2 (0.9) [0.9 to 1.4] | 0.2 (0.0) [0.0 to 0.5]
Statistical Analysis 1: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.4832, Mixed Models Analysis; LSM difference = -0.1, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 2: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.6553, Mixed Models Analysis; LSM difference = -0.1, 95% CI 2-sided [-0.3 to 0.2]
Statistical Analysis 3: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; LSM difference = 0.0, 95% CI 2-sided [-0.2 to 0.3]
Statistical Analysis 4: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.3, 95% CI 2-sided [-1.5 to -1.1]
Statistical Analysis 5: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -2.0, 95% CI 2-sided [-2.2 to -1.7]
Statistical Analysis 6: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 4]; Test type: Superiority; LSM difference = -0.7, 95% CI 2-sided [-0.9 to -0.4]
Statistical Analysis 7: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.3, 95% CI 2-sided [-1.7 to -1.0]
Statistical Analysis 8: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -2.2, 95% CI 2-sided [-2.5 to -1.8]
Statistical Analysis 9: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; LSM difference = -0.8, 95% CI 2-sided [-1.1 to -0.5]
Statistical Analysis 10: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.0, 95% CI 2-sided [-1.4 to -0.6]
Statistical Analysis 11: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.8, 95% CI 2-sided [-2.2 to -1.4]
Statistical Analysis 12: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 10]; Test type: Superiority; LSM difference = -0.8, 95% CI 2-sided [-1.1 to -0.5]
Statistical Analysis 13: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; p = 0.0020, Mixed Models Analysis; LSM difference = -0.8, 95% CI 2-sided [-1.2 to -0.3]
Statistical Analysis 14: Comparison: PF-04965842 200 mg OL to Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSM difference = -1.7, 95% CI 2-sided [-2.2 to -1.2]
Statistical Analysis 15: Comparison: PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB vs PF-04965842 200 mg OL to PF-04965842 200 mg DB; [analysis description as in outcome 22, analysis 13]; Test type: Superiority; LSM difference = -0.9, 95% CI 2-sided [-1.3 to -0.6]

ADVERSE EVENTS:
Time Frame: From screening up to 28 days after last dose of study treatment (maximum up to Week 56)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all participants who received at least 1 dose of study medication.
Groups:
- PF-04965842 200 mg OL: Participants received 12 weeks induction treatment of 200 mg oral tablets (each tablet of 100 mg) PF-04965842 QD during an OL run-in period. Responders at the end of the 12-week open-label run-in period entered the 40 weeks, DB, maintenance treatment period. Responder criteria was defined as a) achieving an IGA of clear (0) or almost clear (1) (on a 5-point scale), b) a reduction from IGA baseline of >= 2 points, and c) reaching an EASI-75 response compared to baseline score. Baseline score was the IGA score and EASI score obtained prior to dosing on Day 1. Non-responders had a choice to enroll into the PF-04965842 LTE study B7451015 (NCT03422822) otherwise, they were permanently discontinued from treatment and were followed-up for 4-week in this study.
- PF-04965842 200 mg OL to Placebo DB: Responders from open-label run-in period received two placebo tablets matched to PF-04965842 orally QD during DB period for up to 40 weeks. Participants who met the protocol defined flare criteria entered in open-label rescue period (RP). Flare was define as a loss of at least 50 percent (%) of the EASI response at Week 12 and had an IGA score of 2 or higher. Participants who did not met the flare criteria had a choice to enroll into the LTE study, otherwise they were permanently discontinued from treatment and were followed-up for 4-week in this study.
Arm/Group | PF-04965842 200 mg OL | PF-04965842 200 mg OL to Placebo DB | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB | PF-04965842 200 mg OL to PF-04965842 200 mg DB | PF-04965842 200 mg Rescue Period
All-Cause Mortality (participants affected / at risk) | 1/1233 | 0/267 | 0/265 | 0/266 | 0/351
Serious Adverse Events (participants affected / at risk) | 20/1233 | 3/267 | 9/265 | 14/266 | 4/351
Other Adverse Events (participants affected / at risk) | 482/1233 | 158/267 | 130/265 | 152/266 | 75/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04965842 200 mg OL (N=1233) | PF-04965842 200 mg OL to Placebo DB (N=267) | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB (N=265) | PF-04965842 200 mg OL to PF-04965842 200 mg DB (N=266) | PF-04965842 200 mg Rescue Period (N=351)
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Eczema herpeticum (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hepatitis E (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04965842 200 mg OL (N=1233) | PF-04965842 200 mg OL to Placebo DB (N=267) | PF-04965842 200 mg OL to PF-04965842 100 mg+Placebo DB (N=265) | PF-04965842 200 mg OL to PF-04965842 200 mg DB (N=266) | PF-04965842 200 mg Rescue Period (N=351)
Blood creatine phosphokinase increased (Investigations) | 43 | 11 | 18 | 25 | 9
Headache (Nervous system disorders) | 119 | 31 | 24 | 31 | 12
Nausea (Gastrointestinal disorders) | 199 | 44 | 35 | 49 | 12
Acne (Skin and subcutaneous tissue disorders) | 68 | 19 | 22 | 31 | 7
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 45 | 88 | 56 | 36 | 13
Nasopharyngitis (Infections and infestations) | 77 | 26 | 27 | 28 | 17
Upper respiratory tract infection (Infections and infestations) | 63 | 26 | 22 | 22 | 21
Vomiting (Gastrointestinal disorders) | 42 | 7 | 12 | 15 | 4

LIMITATIONS AND CAVEATS:
For outcome measure, Time to loss of response, the data collection window was extended for 45 days beyond the scheduled visit due to COVID 19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT03627767/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT03627767/SAP_001.pdf